CLINICAL TRIAL: NCT00549679
Title: A Randomised, Double-blind, Placebo-controlled Study to Investigate the Safety and Tolerability of Inhaled GSK256066 in Mild to Moderate COPD Patients
Brief Title: Study To Evaluate Safety And Tolerability Of GSK256066 In Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IPC101939
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease (COPD); COPD; Repeat Dose; GSK256066
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — 6-((3-((dimethylamino)carbonyl)phenyl)sulfonyl)-8-methyl-4-((3-methyloxyphenyl)amino)-3-quinolinecarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 25 mcg (Experimental): 25 microgram inhaled once daily
  Interventions: Drug: GSK256066
- 87.5 mcg (Experimental): 87.5 microgram inhaled once daily
  Interventions: Drug: GSK256066
- Placebo (Placebo Comparator): Placebo inhaled once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK256066 — PDE4 inhibitor
  Arms: 25 mcg; 87.5 mcg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and tolerability of the cfor the first time in mild to moderate COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Male adults or female adults of non-childbearing potential who are between 40 and 75 years of age (inclusive).
* Subjects with a clinical diagnosis of COPD in accordance with the European Respiratory Society Consensus Statement and subjects categorised with moderate COPD as defined by the GOLD guidelines of 2006 [GOLD, 2006]
* Subjects with a cigarette smoking history of ≥ 10 pack years (1 pack year = 20 cigarettes smoked per day for 1 year or the equivalent). Both current and former smokers are eligible to be enrolled. A former smoker is defined as a subject who has not smoked for ≥6 months at Visit 1.
* Subjects with a post-bronchodilator FEV1 to FVC ratio (FEV1/FVC) < 0.7 at Visit 1. Subjects will be assessed 30 (± 5) minutes after receiving salbutamol 400 μg.
* Subjects with a post-bronchodilator FEV1 ≥ 50% and < 80% of predicted normal for height, age and sex at Visit 1. Subjects will be assessed 30 (± 5) minutes after receiving salbutamol 400 μg.
* Subjects with a normal echocardiogram at screening, as defined by the absence of clinically significant wall motion, chamber size or valvular abnormalities
* The subject must be capable of giving informed consent and can comply with the study requirements and timetable.

Exclusion Criteria:

* Women who are pre-menopausal and of child-bearing potential.
* Subjects weighing less than 50 kilograms (kg).
* Subjects who are obese defined as having a body mass index (BMI) > 30.
* Subjects with a current diagnosis of asthma.
* Subjects who have required hospitalisation or treatment with oral corticosteroids and/or antibiotic therapy for acute worsening of COPD or lower respiratory tract infection in the 6 weeks prior to Screening.
* Subjects who have received treatment with oral, intravenous, topical or intra-articular corticosteroids within 6 weeks of Screening or thereafter
* Subjects with active tuberculosis, sarcoidosis or clinically overt bronchiectasis.
* Subjects with a history of any type of malignancy with the exception of successfully treated squamous cell cancer of the skin.
* Subjects with rheumatoid arthritis, connective tissue disorders and other conditions known to be associated with chronic inflammation (e.g. Inflammatory Bowel Disease).
* Subjects with chronic infections (lasting longer than 6 months) such as gingivitis, periodontitis, prostatitis, gastritis, and urinary tract infections.
* Subjects with any acute infection, sinus symptoms, or significant trauma (burns, fractures).
* Subjects with clinically significant renal disease, diabetes mellitus/metabolic syndrome, hypertension or any other clinically significant cardiovascular, neurological, endocrine, or haematological abnormalities that are uncontrolled on permitted therapy.
* Subjects who have participated in any GSK study/studies involving administration of COA.
* The subject has a screening ECG parameters outside of ranges specified in protocol.
* Subjects with hypoxaemia
* Risk factors for human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C infection at Screening (Visit 1).
* Subjects who have undergone surgery including lung volume reduction surgery in the last six months or have conditions that prevent them from performing spirometry.
* Subjects with a history (or suspected history) of alcohol misuse or any other recreational substance abuse.
* Subjects who require treatment with any of the following from the start of the run-in period (Day -14) until the end of the treatment phase:
* Inhaled corticosteroids
* Inhaled cromolyn sodium or nedocromil
* Xanthines (theophylline preparations).
* Leukotriene modifiers
* Tiotropium
* Long-acting inhaled beta2-agonists (salmeterol, formoterol)
* Oral beta2-agonists
* Subjects who are unable to abstain from other courses of medication during the run in phase including non-steroidal anti-inflammatory drugs (NSAIDs), anti-depressant drugs, anti-histamines, anti-rhinitis or hay fever medication, other than short acting inhaled beta-agonists, ipratropium bromide and paracetamol (up to 4 g per day) for the treatment of minor ailments (eg headache) from 48h before the first dose until the follow-up visit. Subjects requiring medication between dosing and follow up may be excluded at the principal investigators discretion.
* Subjects with any known hypersensitivity to salbutamol or ipratropium bromide.
* Subjects who are participating or plan to participate in the active phase of a pulmonary rehabilitation programme during the study.
* Subjects who have received an investigational drug within 30 days or within five drug half-lives of the investigational drug (whichever is longer).
* Subjects with any clinically relevant abnormality detected by the assessments at Screening.
* Subjects who have experienced an exacerbation during the run-in period requiring treatment with oral corticosteroids and/or macrolide antibiotics and/or hospitalisation.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2007-10-04; Primary Completion 2008-12-15 (Actual); Study Completion 2008-12-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to follow up (approximately 56 days)
  An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention.
Change from Baseline (Day 0 [pre-bronchodilator]) in 12-lead electrocardiogram (ECG) findings | Baseline (Day 0 [pre-bronchodilator]) and up to Day 28 (Visit 6b)
  ECG parameters consist of QT interval corrected by Bazett's (QTcB) and Fridericia's (QTcF) formulas, QT interval, QRS duration and PR interval. Baseline was defined as value at Day 0 (pre-bronchodilator). The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline was the mean of the 3 pre-salbutamol measurements at Day 0. It was assessed on Baseline, Day 1, 7, 14, 15, 21, 27 and 28. Post Baseline, ECG was performed 1-2 hours post dose.
Change from Baseline (Day 0 [pre-bronchodilator]) in 12-lead electrocardiogram (ECG) findings-ventricular rate | Baseline (Day 0 [pre-bronchodilator]) and up to Day 28 (Visit 6b)
  ECG parameters consist of ventricular rate. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline was the mean of the 3 pre-salbutamol measurements at Day 0. It was as/sessed on Baseline, Day 1, 7, 14, 15, 21, 27 and 28. Post Baseline, ECG was performed 1-2 hours post dose.
Number of participants with abnormal (potential clinical importance [PCI]) systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate (HR) | Up to Day 27 (Visit 6a)
  The PCI range for SBP was < 85 and > 160 millimeters of mercury (mmHg), DBP was < 45 and > 100 mmHg and for HR < 40 and > 110 beats per minute. It was assessed on Baseline (pre-bronchodilator), Day 14 and 27. Data for SBP high, SBP low, DBP high, DBP low, HR high and HR low is presented.
Number of participants with abnormal (PCI) clinical chemistry | Up to Day 42 (follow up visit)
  Clinical chemistry included: albumin, bicarbonate, alanine aminotransferase (ALT), albumin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), blood urea, creatinine, magnesium, sodium, potassium, chloride, glucose, total bilirubin, direct bilirubin, indirect bilirubin, total protein, gamma glutamyltransferase (GGT), calcium, creatinine kinase, creatine kinase-MB, creatinine clearance (estimated; male and female), lactate dehydragenase, and troponin, triglycerides. Data for abnormal parameters (above and below range) is provided. It was assessed on Baseline (Day -3), Day 14, 28 and on follow up visit (Day 42). Data for only abnormal observations is presented.
Number of participants with abnormal (PCI) hematology | Up to Day 42 (follow up visit)
  Hematology included: haemoglobin, haematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red blood cell (RBC) indices, white blood cell (WBC), basophils, eosinophils, lymphocytes, monocytes, neutrophils and platelet count. Data for abnormal parameters (above and below range) is provided. It was assessed on Baseline (Day -3), Day 14, 28 and on follow up visit (Day 42). Data for only abnormal observations is presented.
Number of participants with abnormal urinalysis | Up to Day 56 (Visit follow up)
  Abnormal urinalysis data for RBC in urine and haematuria presented. Data for abnormal parameters (above and below range) is provided. It was assessed on Baseline (Day -3), Day 7, 14, 21, 28 and on follow up visit (Day 42). Data for only abnormal observations is presented.
Change from Baseline (Day 0) in lung function parameters: forced expiratory volume in one second (FEV1) and forced vital capacity (FVC) | Baseline (Day 0) and up to Day 27 (Visit 6a)
  The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline value defined as the value on Day 0. It was assessed on Baseline (Day 0), Day 14 and 27. Spirometry tests was performed before and 30 minutes after dosing with salbutamol (bronchodilator) on Day 0 and before dosing with GSK256066. As they were analyzed separately, there were two Baselines for these tests, 'pre bronchodilator Baseline' and 'post bronchodilator Baseline'. Smoking and short acting bronchodilators were avoided 6 hour prior to administration of the salbutamol. Observations with best test review (BTR) grading of 'not acceptable' were excluded.
Number of participants with abnormal Holter interpretations | Up to Day 27 (Visit 6a)
  Holter parameters were derived by visit over the 24 hour period as: maximum HR over 24 hours was the maximum HR of all time slices and mean HR over 24 hours was the mean HR of all time slices, weighted by the time length of each slice. The total number of ventricular runs and the number of supraventricular runs over 24 hours were derived by summing each count across all time slices. Data for normal, abnormal: not clinically significant and abnormal: clinically significant is presented. It was assessed on Baseline (Day 0), Day 14and 27. Data for normal, abnormal: clinically significant and abnormal: clinically not significant presented.
Number of participants who withdrawn for exacerbations of chronic obstructive pulmonary disease (COPD) | Up to Day 27 (Visit 6a)
  An exacerbation of COPD was defined as worsening of COPD symptoms requiring changes to normal treatment including antimicrobial therapy, short courses of oral steroids and other bronchodilator therapy. If clinically indicated, short-term treatment with antibiotics could be prescribed for the exacerbation. Any participants requiring treatment with inhaled or oral corticosteroids or admission to hospital were withdrawn from the study.

SECONDARY OUTCOMES:
Plasma concentrations of GSK256066 and active metabolite GSK614917 and derived pharmacokinetic parameters: area under the plasma drug concentration versus time curve (AUC0-last) | Pre-dose and at 15, 30 minutes, 1, 2, 3, 4, 6, 8, 10 and 24 hour post dosing at Baseline (Visit 2a) and Days 14 and 27 (Visits 4a and 6a)
  AUC0-last determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. AUC0-last for GSK256066 is presented. As GSK614917 concentrations were generally non-quantifiable, no summary statistics were derived for GSK614917 pharmacokinetic parameters due to the large number of missing values resulting from non-quantifiable concentration-time data. AUC(0-t) imputed with half lowest observed AUC(0-t) (half of 1.28 hour×picogram/ milliliters [mL]).
Plasma concentrations of GSK256066 and active metabolite GSK614917 and derived pharmacokinetic parameters: maximum observed plasma drug concentration (Cmax) | Pre-dose and at 15, 30 minutes, 1, 2, 3, 4, 6, 8, 10 and 24 hour post dosing at Baseline (Visit 2a) and Days 14 and 27 (Visits 4a and 6a)
  The first occurrence of the maximum observed concentration determined directly from the raw concentration-time data. Cmax for GSK256066 is presented. As GSK614917 concentrations were generally non-quantifiable, no summary statistics were derived for GSK614917 pharmacokinetic parameters due to the large number of missing values resulting from non-quantifiable concentration-time data. One pre-dose GSK614917 concentration at the Baseline visit which was >5% of the corresponding Cmax was excluded from the pharmacokinetic analysis. Cmax imputed with half lower limit of quantification (LLQ; half of 5 picogram/mL).
Plasma concentrations of GSK256066 and GSK614917 and derived pharmacokinetic parameters: time to maximum observed plasma drug concentration (tmax) | Pre-dose and at 15, 30 minutes, 1, 2, 3, 4, 6, 8, 10 and 24 hour post dosing at Baseline (Visit 2a) and Days 14 and 27 (Visits 4a and 6a)
  The tmax was the time at which Cmax was observed. Tmax was determined directly from the raw concentration-time data. Pharmacokinetic data of GSK256066 is presented. As GSK614917 concentrations were generally non-quantifiable, no summary statistics were derived for GSK614917 pharmacokinetic parameters due to the large number of missing values resulting from non-quantifiable concentration-time data.
Change from Baseline (Day -3) total cell number (cells/mL) in induced sputum | Baseline (Day -3) and Day 28 (Visit 6b)
  Sputum was performed using ipratropium bromide. Participants must fast for 2 hour prior to the sputum induction (only water was allowed) and on Day 28 (Visit 6b), it was performed 2-4 hours after the final dose of study medication. One participant had a total number of neutrophil cell/ mLs count of 0 which was imputed to 1. Data for adjusted geometric means of macrophages, neutrophils cells per mLs and total leukocyte count is presented as geometric mean. The change from Baseline was calculated by subtracting the Baseline values from the Day 28 values. Baseline was defined as the value at Day -3. Total number of cells per mL was calculated by percentage of cells divided by 100 multiplied by total leukocyte count. It was assessed on Baseline and Day 28.
Change from Baseline (Day -3) in neutrophils and macrophages as a percentage of total cells in induced sputum | Baseline (Day -3) and Day 28 (Visit 6b)
  Sputum was performed using ipratropium bromide. Participants must fast for 2 hour prior to the sputum induction (only water was allowed) and on Day 28 (Visit 6b), it was performed 2-4 hours after the final dose of study medication. One participant had a total number of neutrophil cell/ mLs count of 0 which was imputed to 1. Data for adjusted means of percentage of total cells macrophages and neutrophils is presented as least square mean. The change from Baseline was calculated by subtracting the Baseline values from the Day 28 values. Baseline was defined as the value at Day -3. Percentage cells was calculated by absolute cell count divided by total non squamous cell count multiplied by 100. It was assessed on Baseline and Day 28.
Summary of mean lymphocytes, bronchial epithelial cells and eosinophils as a percentage of total cells in induced sputum | Up to Day 28 (Visit 6b)
  Sputum was performed using ipratropium bromide. Participants must fast for 2 hour prior to the sputum induction (only water was allowed) and on Day 28 (Visit 6b), it was performed 2-4 hours after the final dose of study medication. Data for adjusted means of percentage of total cells macrophages and neutrophils is presented as geometric mean. The change from Baseline was calculated by subtracting the Baseline values from the Day 28 values. Baseline was defined as the value at Day -3. Percentage cells was calculated by absolute cell count divided by total non squamous cell count multiplied by 100. It was assessed on Baseline and Day 28.
Absolute numbers of leukocytes, neutrophils and macrophages in induced sputum | Up to Day 28 (Visit 6b)
  Sputum was performed using ipratropium bromide. Participants must fast for 2 hour prior to the sputum induction (only water was allowed) and on Day 28 (Visit 6b), it was performed 2-4 hours after the final dose of study medication. One participant had a total number of neutrophil cell/ mLs count of 0 which was imputed to 1. Total number of cells per mL was calculated by percentage of cells divided by 100 multiplied by total leukocyte count. It was assessed on Baseline and Day 28. One participant had a total number of neutrophil cell/ mLs count of 0 which was imputed to 1.
Absolute numbers of bronchial epithelial cells, lymphocytes and eosinophils in induced sputum | Up to Day 28 (Visit 6b)
  Sputum was performed using ipratropium bromide. Participants must fast for 2 hour prior to the sputum induction (only water was allowed) and on Day 28 (Visit 6b), it was performed 2-4 hours after the final dose of study medication. One participant had a total number of neutrophil cell/ mL count of 0 which was imputed to 1. Total number of cells per mL was calculated by percentage of cells divided by 100 multiplied by total leukocyte count. It was assessed on Baseline and Day 28.
Summary of concentration of total protein in induced sputum supernatant | Up to Day 28 (Visit 6b)
  Sputum was performed using ipratropium bromide. Participants must fast for 2 hour prior to the sputum induction (only water was allowed) and on Day 28 (Visit 6b), it was performed 2-4 hours after the final dose of study medication. It was assessed on Baseline and Day 28. Values below LLQ or above upper limit of quantification (ULQ) was imputed to half the LLQ or ULQ, LLQs: total protein: 62.5 µg/mL and ULQ: total protein: 400 µg/mL. Adjusted mean values for current smokers and former smokers is presented as least square mean.
The concentration of inflammatory biomarkers in induced sputum supernatant: interleukin (IL) 8 | Up to Day 28 (Visit 6b)
  Sputum was performed using ipratropium bromide. Participants must fast for 2 hour prior to the sputum induction (only water was allowed) and on Day 28 (Visit 6b), it was performed 2-4 hours after the final dose of study medication. It was assessed on Baseline and Day 28. Values below LLQ or above ULQ was imputed to half the LLQ or ULQ, LLQs: IL8: 70000 picograms/mL and ULQ: IL8: 360000 picograms/mL.
The concentration of inflammatory biomarkers in induced sputum supernatant: myeloperoxidase (MPO) | Up to Day 28 (Visit 6b)
  Sputum was performed using ipratropium bromide. Participants must fast for 2 hour prior to the sputum induction (only water was allowed) and on Day 28 (Visit 6b), it was performed 2-4 hours after the final dose of study medication. It was assessed on Baseline and Day 28. Values below LLQ or above ULQ was imputed to half the LLQ or ULQ, LLQs: MPO: 90 nanograms/mL and ULQ: IL8: 5000 nanograms/mL.
Summary of messenger ribonucleic acid (mRNA) and/or protein in induced sputum of established and exploratory markers of inflammation: IL-6, IL-1 beta and IL-8 | Day 28 (Visit 6b)
  Sputum was performed using ipratropium bromide. Participants must fast for 2 hour prior to the sputum induction (only water was allowed) and on Day 28 (Visit 6b), it was performed 2-4 hours after the final dose of study medication. It was assessed on Baseline and Day 28. Data for adjusted mean is presented as least square mean.
Summary of mRNA and/or protein in induced sputum of established and exploratory pharmacodynamic markers: Phosphodiesterase-4 B (PDE4B), SNF1 like kinase (SNF1LK) | Up to Day 28 (Visit 6b)
  Sputum was performed using ipratropium bromide. Participants must fast for 2 hour prior to the sputum induction (only water was allowed) and on Day 28 (Visit 6b), it was performed 2-4 hours after the final dose of study medication. It was assessed on Baseline and Day 28.
Summary of lung function parameters (pre and post-bronchodilator): mean spirometry measures FEV1 and FVC | Up to Day 27 (Visit 6a)
  Spirometry tests was performed before and 30 minutes after dosing with salbutamol (bronchodilator) on Day 0 and before dosing with GSK256066. As they were analyzed separately, there were two Baselines for these tests, 'pre bronchodilator Baseline' and 'post bronchodilator Baseline'. Smoking and short acting bronchodilators were avoided 6 hour prior to administration of the salbutamol. It was assessed on Baseline (Day 0), Day 14 and 27. Observations with BTR grading of 'not acceptable' were excluded.
Summary of lung function parameters (pre and post-bronchodilator): plethysmography measures: inspiratory capacity (IC), residual volume (RV), total lung capacity (TLC), slow vital capacity (SVC) and thoracic gas volume (TGV) | Up to Day 27 (Visit 6a)
  Plethysmography procedures was performed 30 minutes after dosing with salbutamol and prior to dosing with GSK256066. Participants were resting in the body box for at least 1 minute prior to any assessments. Smoking and short acting bronchodilators should be avoided 6 hour prior to administration of the salbutamol. It was assessed on Baseline (Day 0) and 27. Data for adjusted mean is presented as least square mean.
Summary of lung function parameters (pre and post-bronchodilator): plethysmography measures: plus airway resistance (Raw) | Up to Day 27 (Visit 6a)
  Plethysmography procedures was performed 30 minutes after dosing with salbutamol and prior to dosing with GSK256066. Participants were resting in the body box for at least 1 minute prior to any assessments. Smoking and short acting bronchodilators should be avoided 6 hour prior to administration of the salbutamol. It was assessed on Baseline (Day 0) and 27. Data for adjusted mean is presented as least square mean.
Summary of lung function parameters (pre and post-bronchodilator): plethysmography measures: specific airway conductance (sGaw) | Up to Day 27 (Visit 6a)
  Plethysmography procedures was performed 30 minutes after dosing with salbutamol and prior to dosing with GSK256066. Participants were resting in the body box for at least 1 minute prior to any assessments. Smoking and short acting bronchodilators should be avoided 6 hour prior to administration of the salbutamol. It was assessed on Baseline (Day 0) and 27. Data for adjusted mean is presented as least square mean.
Summary of lung function parameters (pre and post-bronchodilator): impulse oscillometry (IOS): total resistance (R5) and large airway resistance (R25); low frequence reactance (X5) | Up to Day 27 (Visit 6a)
  IOS tests were performed prior to other measurements of pulmonary function to avoid any influence of forced expiratory manoeuvres on airway function during resting breathing. IOS test was performed before and 30 minutes after dosing with salbutamol and before dosing with GSK256066. Smoking and short acting bronchodilators should be avoided 6 hour prior to administration of the salbutamol. It was assessed on Baseline (Day 0) and 27. Observations with BTR grading of 'not acceptable' were excluded. Data for adjusted mean is presented as least square mean.
Summary of lung function parameters (pre and post-bronchodilator): IOS-resonant frequency (RF) | Up to Day 27 (Visit 6a)
  IOS tests were performed prior to other measurements of pulmonary function to avoid any influence of forced expiratory manoeuvres on airway function during resting breathing. IOS test was performed before and 30 minutes after dosing with salbutamol and before dosing with GSK256066. Smoking and short acting bronchodilators should be avoided 6 hour prior to administration of the salbutamol. It was assessed on Baseline (Day 0) and 27. Observations with BTR grading of 'not acceptable' were excluded. Data for adjusted mean is presented as least square mean.
Summary of lung function parameters (pre and post-bronchodilator): impulse oscillometry (IOS): peripheral resistance (R5-R15) and R15 | Up to Day 27 (Visit 6a)
  IOS tests were performed prior to other measurements of pulmonary function to avoid any influence of forced expiratory manoeuvres on airway function during resting breathing. IOS test was performed before and 30 minutes after dosing with salbutamol and before dosing with GSK256066. Smoking and short acting bronchodilators should be avoided 6 hour prior to administration of the salbutamol. It was assessed on Baseline (Day 0) and 27. Observations with BTR grading of 'not acceptable' were excluded. The parameter 'R5-R15' was derived by subtracting R15 from R5 for each subject at each time point.
Summary of lung function parameters (pre and post-bronchodilator): IOS-low frequence reactance area (AX) | Up to Day 27 (Visit 6a)
  IOS tests were performed prior to other measurements of pulmonary function to avoid any influence of forced expiratory manoeuvres on airway function during resting breathing. IOS test was performed before and 30 minutes after dosing with salbutamol and before dosing with GSK256066. Smoking and short acting bronchodilators should be avoided 6 hour prior to administration of the salbutamol. It was assessed on Baseline (Day 0) and 27. Observations with BTR grading of 'not acceptable' were excluded.
The concentration of serum inflammatory biomarkers: fibrinogen | Up to Day 28 (Visit 6b)
  Blood samples were collected to determine serum concentrations of inflammation biomarkers such as fibrinogen, tumour necrosis factor (TNF)-alpha, soluble TNF receptors (sTNF-Rs), IL-8, IL-6, IL-1-beta using an appropriately validated assay including ELISA and multiplex analysis. TNFα, sTNF-Rs, IL-8, IL-6 and IL-1-beta data were not collected. Values below LLQ or above ULQ have been imputed to half the LLQ or ULQ. LLQ for fibrinogen-0.4 grams per liter and ULQs for fibrinogen-14 grams per liter. Data for adjusted mean is presented as least square mean.
The concentration of serum inflammatory biomarkers: surfactant protein-D (SP-D) | Up to Day 28 (Visit 6b)
  Blood samples were collected to determine serum concentrations of inflammation biomarkers such as fibrinogen, tumour necrosis factor-alpha (TNF-alpha), sTNF-Rs, IL-8, IL-6, IL-1-beta using an appropriately validated assay including ELISA and multiplex analysis. TNFα, sTNF-Rs, IL-8, IL-6 and IL-1-beta data were not collected. Surfactant protein D (SP-D) was collected. Values below LLQ or above ULQ have been imputed to half the LLQ or ULQ. LLQ for SP-D-7.8 nanograms per mL and ULQs for SP-D-2000 nanograms per mL. Data for adjusted mean is presented as least square mean.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- GSK Investigational Site, Tallinn, Estonia
- GSK Investigational Site, Tampere, Finland
- Germany (3):
  - GSK Investigational Site, Gauting, Bavaria
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Netherlands (3):
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Horn
  - GSK Investigational Site, Veldhoven
- Russia (4):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Yaroslavl
- Slovakia (3):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Martin

REFERENCES:
- [Derived] Watz H, Mistry SJ, Lazaar AL; IPC101939 investigators. Safety and tolerability of the inhaled phosphodiesterase 4 inhibitor GSK256066 in moderate COPD. Pulm Pharmacol Ther. 2013 Oct;26(5):588-95. doi: 10.1016/j.pupt.2013.05.004. Epub 2013 May 21. PMID 23701917